CLINICAL TRIAL: NCT00575614
Title: Study to Evaluate the Effect of a 1 mg o.d. Dose of Prucalopride in Patients With Chronic Idiopathic Constipation
Brief Title: Prucalopride in Patients With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBR-4
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-12

CONDITIONS: Constipation
Keywords: Constipation; Prucalopride; Ano-rectal physiology; Oro-caecal transit time; QOL
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: prucalopride
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prucalopride — 1 mg o.d.
  Other Names: Resolor
  Arms: 1
Drug: placebo — o.d.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in the treatment of chronic idiopathic constipation.

Hypothesis:

Prucalopride given at a dose of 1 mg o.d. for 4 weeks to female patients with chronic constipation shows a favourable effect on most of the efficacy parameters assessed in this trial. This dosage can be considered safe and generally well-tolerated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, phase II trial set up to investigate the efficacy, safety and physiological effects of prucalopride 1 mg administered o.d. for 4 weeks to female patients with chronic idiopathic constipation. The primary objective of this trial was to assess the effect of prucalopride 1 mg on whole gut transit (measured as changes from baseline in total number of markers).

ELIGIBILITY:
Inclusion Criteria:

* female subjects of 18 years or over;
* history of chronic constipation during at least 6 months before selection, characterized by either two or fewer spontaneous (ie, without using laxatives) bowel movements in a week or straining at defaecation at least a quarter of the time;
* written informed consent;
* within 20% of her body weight as specified in the Metropolitan Life Insurance Company's 1983 Height and Weight Table2;
* healthy on the basis of a pre-trial physical examination, medical history, anamnesis,electrocardiogram and the results of biochemistry, haematology and urinalysis, carried out within 3 weeks of randomization. If the results of the laboratory tests were not within the reference ranges, the subject could only be included on condition that the investigator did not judge the deviations to be clinically relevant.

Exclusion Criteria:

* use of disallowed concomitant medication;
* subjects who had undergone surgery for their constipation;
* subjects with faecal impaction;
* subjects suffering from different types or causes of constipation other than idiopathic constipation, ie, presence of secondary causes, eg, endocrine disorders, metabolic disorders, neurologic disorders;
* subjects with a megacolon/megarectum;
* subjects with external rectal prolapse;
* history of previous abdominal surgery (other than hysterectomy, surgery for Meckel's diverticle, appendectomy, cholecystectomy, inguinal hernia repair, splenectomy, nephrectomy or fundoplication) thought to be the primary cause of constipation;
* known or suspected organic disorders of the large bowel, ie, obstruction, carcinoma or inflammatory bowel disease. If complaints of constipation were of recent onset, ie, had been present for less than one year, and the subject was 40 years or older, results of a Ba-enema or of colonoscopic examination were required;
* subjects with solitary rectal ulcer (this had to be excluded by rigid sigmoidoscopic examination at the first visit);
* subjects with active proctological conditions thought to be responsible for the constipation;
* subjects with known illnesses or conditions such as: severe cardiovascular or lung disease, neurologic or psychiatric disorders (including substance abuse/dependence, but with the exception of nicotine), alcoholism, cancer or AIDS and other gastrointestinal or endocrine disorders;
* subjects receiving, or who had received, care for an eating disorder;
* subjects with impaired renal function;
* subjects with a serum amylase, a serum glutamic-oxaloacetic transaminase (SGOT), or a serum glutamic-pyruvic transaminase (SGPT) concentration of > 2 times the normal limit;
* pregnancy or wish to become pregnant in the course of the trial. Lack of an acceptable birth control method;
* breast-feeding;
* subjects who had received an investigational drug in the 30 days preceding the trial;
* subjects who were unable or unwilling to return for required follow-up visits;
* subjects whose reliability and physical state would prevent proper evaluation of a drug trial;
* history or suspicion of alcohol or drug abuse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 1997-04; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Whole gut transit | 4 weeks

SECONDARY OUTCOMES:
Ano-rectal physiology | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kamm, MD, Principal Investigator — Northwick Park Hospital

REFERENCES:
- [Result] Emmanuel AV, Roy AJ, Nicholls TJ, Kamm MA. Prucalopride, a systemic enterokinetic, for the treatment of constipation. Aliment Pharmacol Ther. 2002 Jul;16(7):1347-56. doi: 10.1046/j.1365-2036.2002.01272.x. PMID 12144586